CLINICAL TRIAL: NCT06801444
Title: Comparison of Intr-operative Neuromonitoring Technique in Trans-oral Endoscopic Thyroidectomy Vestibular Approach
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yih-Huei Uen, Attending physician, China Medical University Hospital
Other Study IDs: CMUH113-REC3-170
Record Dates: First submitted 2025-01-07; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Transoral endoscopic thyroidectomy vestibular approach (TOETVA) has the advantage of scarless cosmesis but has limitations of recurrent laryngeal nerve (RLN) palsy. Intermittent intraoperative neuromonitoring (I-IONM) techniques have been utilized during TOETVA to identify and map RLN to prevent RLN injury. However, the insult may still occur between two neural stimulations. Continuous intraoperative neuromonitoring (C-IONM) has been used in TOETVA to persistent stimulation of RLN. but only in our hospital. This rare use may be related to technical challenges. Recently, we successfully developed a novel technique of percutaneous C-IONM using an external fixator to secure the stimulation probe to steadily monitor the real-time functional status of RLN during the TOETVA. In this retrospective study, 304 patients undergone TOETVA were enrolled and divided according to the usage of IONM techniques into percutaneous or peroral intermittent and continuous groups. Patient's age, sex, BMI, thyroid disease, operation time, EMG signal and RLN palsy rate were compared to verified the feasibility, safety, and effectiveness of different IONM techniques. We hypothesized percutaneous C-IONM has the superiority in early detection of RLN injury and reducing of RLN palsy in TOETVA.

ELIGIBILITY:
Inclusion Criteria: Benign solitary or multiple thyroid nodules, follicular lesions (the largest diameter <6.0 cm), and early papillary thyroid carcinoma (<1 cm in diameter, without cervical lymphadenopathy)

Exclusion Criteria: History of thyroid surgery, neck radiotherapy, and recurrent laryngeal nerve paralysis; intraoperative conversion to conventional thyroidectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing transoral vestibular endoscopic total thyroidectomy.
Sampling Method: Probability Sample
Enrollment: 304 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
Electrode set up time refers to the time (min) from endoscopic or percutaneous insertion of electrode to functional set up of neural stimulation | through study completion, an average of one year
Operative time refers to the time (min) from incision wound making to complete wound closure | through study completion, an average of one year
Times of intraoperative displacement of stimulator electrode refers to total number of electrode displacement resulting in abnormal EMG signal | through study completion, an average of one year
Stimulation intensity refers to the level (mA) of stimulation current used | through study completion, an average of one year
Recurrent laryngeal nerve palsy refers to the presence of fixed or immobile vocal cord in laryngeal scopic examination | through study completion, an average of one year
EMG signals refers to the amplitude (μV) and latency (ms) of biphasic EMG wave recorded from vocal cord with neural stimulation | through study completion, an average of one year

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Chen HK, Chen CL, Wen KS, Lin YF, Lin KY, Uen YH. Application of transoral continuous intraoperative neuromonitoring in natural orifice transluminal endoscopic surgery for thyroid disease: a preliminary study. Surg Endosc. 2018 Jan;32(1):517-525. doi: 10.1007/s00464-017-5656-0. Epub 2017 Jun 22. PMID 28643050
- [Background] Lamade W, Ulmer C, Seimer A, Molnar V, Meyding-Lamade U, Thon KP, Koch KP. A new system for continuous recurrent laryngeal nerve monitoring. Minim Invasive Ther Allied Technol. 2007;16(3):149-54. doi: 10.1080/13645700701383241. PMID 17573619
- [Background] Schneider R, Machens A, Sekulla C, Lorenz K, Elwerr M, Dralle H. Superiority of continuous over intermittent intraoperative nerve monitoring in preventing vocal cord palsy. Br J Surg. 2021 May 27;108(5):566-573. doi: 10.1002/bjs.11901. PMID 34043775
- [Background] Lombardi CP, De Waure C, Mariani M, Carnassale G, D'Amore A, Traini E, De Crea C, Raffaelli M, Damiani G. Efficacy of continuous neuromonitoring in thyroid surgery: preliminary report of a single-center experience. Gland Surg. 2019 Aug;8(4):336-342. doi: 10.21037/gs.2019.08.02. PMID 31538057
- [Background] Schneider R, Randolph G, Dionigi G, Barczynski M, Chiang FY, Triponez F, Vamvakidis K, Brauckhoff K, Musholt TJ, Almquist M, Innaro N, Jimenez-Garcia A, Kraimps JL, Miyauchi A, Wojtczak B, Donatini G, Lombardi D, Muller U, Pezzullo L, Ratia T, Van Slycke S, Nguyen Thanh P, Lorenz K, Sekulla C, Machens A, Dralle H. Prospective study of vocal fold function after loss of the neuromonitoring signal in thyroid surgery: The International Neural Monitoring Study Group's POLT study. Laryngoscope. 2016 May;126(5):1260-6. doi: 10.1002/lary.25807. Epub 2015 Dec 15. PMID 26667156
- [Background] Chiang FY, Lu IC, Chang PY, Sun H, Wang P, Lu XB, Chen HC, Chen HY, Kim HY, Dionigi G, Wu CW. Stimulating dissecting instruments during neuromonitoring of RLN in thyroid surgery. Laryngoscope. 2015 Dec;125(12):2832-7. doi: 10.1002/lary.25251. Epub 2015 Mar 26. PMID 25809677
- [Background] Liu XL, Wu CW, Zhao YS, Wang T, Chen P, Xin JW, Li SJ, Zhang DQ, Zhang G, Fu YT, Zhao LN, Zhou L, Dionigi G, Chiang FY, Sun H. Exclusive real-time monitoring during recurrent laryngeal nerve dissection in conventional monitored thyroidectomy. Kaohsiung J Med Sci. 2016 Mar;32(3):135-41. doi: 10.1016/j.kjms.2016.02.004. Epub 2016 Mar 30. PMID 27106003
- [Background] Tae K. Complications of Transoral Thyroidectomy: Overview and Update. Clin Exp Otorhinolaryngol. 2021 May;14(2):169-178. doi: 10.21053/ceo.2020.02110. Epub 2020 Nov 19. PMID 33211953